CLINICAL TRIAL: NCT06909032
Title: Accelerated Partial Breast Irradiation Using External Beam Volumetric Modulated Arc Therapy (VMAT): a Randomised Non-inferiority Trial of 30 Gy Versus 26 Gy in Five Fractions Investigating Patient-reported Outcomes
Acronym: PUMA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Integrated Community Oncology Network (Other)
Collaborators: Icon Cancer Foundation (ICF) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23.05
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: Partial breast irradiation (PBI); Patient reported outcomes; Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Hypofractionated PBI delivering a total dose of 30 Gy in five consecutive daily fractions. (Active Comparator): PBI will be delivered using a VMAT planning and delivery technique. Prior to treatment patients are required to attend a treatment planning session that will assist with planning the treatment. The planning procedure will take up to approximately 60 minutes and involve a computed-tomography (CT) scan with the patient positioned in the treatment position. Treatment is expected to take around 15 minutes per treatment. The intervention will be prescribed by a radiation oncologist and administered by radiation therapists. During treatment, imaging will be completed to ensure treatment is administered accurately.
  All patients will complete breast cancer related quality of life questionnaires.
  Interventions: Radiation: Accelerated partial breast irradiation
- Arm B: Hypofractionated PBI delivering a total dose of 26 Gy in five consecutive daily fractions. (Active Comparator): The comparator for this study is another dose that is used as standard of care for APBI in Australia and globally.
  Planning and treatment procedures will be same as that for Arm A.
  Interventions: Radiation: Accelerated partial breast irradiation

INTERVENTIONS:
Radiation: Accelerated partial breast irradiation — Accelerated partial breast irradiation (APBI) will be delivered using Volumetric Modulated Arc Therapy (VMAT). Treatment will be started within 12 weeks of breast conserving surgery and within four weeks of randomisation. Treatment will occur in five (5) once-daily sessions and should be completed within seven (7) days of starting radiotherapy. Two total doses of APBI will be compared: 30 Gy and 26 Gy. The aim is to determine whether quality of life is no worse when a higher dose of APBI is used compared to a slightly lower dose of APBI. The results of this study will help to guide doctors choose the best dose of APBI for patients with early breast cancer in the future.

SUMMARY:
For women undergoing radiotherapy following surgery for early-stage breast cancer, breast-related quality of life (BrQoL) is an important consideration. Treating only the part of the breast by radiation where the cancer has been surgically removed (partial breast irradiation or "PBI") rather than the whole breast (whole breast irradiation) can reduce the toxic effects of radiotherapy. This trial aims to evaluate whether there is a difference in patient-reported BrQoL between two total doses of radiation given in five treatments using PBI. If BrQOL for the higher dose of PBI is no worse than the lower dose, using the higher dose would be advised as best practice, given that it is more likely to be more effective in reducing the chance of cancer coming back in the breast than the lower dose.

DETAILED DESCRIPTION:
Single-blind, phase III, multisite, randomised non-inferiority trial. PBI will be planned and treated as per the protocol using VMAT. The prescribed dose will be 30 Gy in 5 daily fractions (Arm A) or 26 Gy in 5 daily fractions (Arm B). Participants will be blinded to their treatment allocation.

Follow-up will be at the following time points:

* Eight weeks following the end of radiation
* Every six months post-randomisation for two years following randomisation
* Three years post-randomisation (final visit)

Assessments to be conducted at each time point are:

* Clinical assessment
* Completion of Patient-Reported Outcome Measures (PROMs)
* Mammogram and ultrasound (baseline and annually)
* Documentation of IBTR - classified as a true recurrence or Elsewhere
* Documentation of any other type of recurrence (regional, distant, opposite breast)

Recruitment is planned for three years with a three-year follow-up period for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged greater than or equal to 50 years old
* Histologically confirmed Infiltrating ductal carcinoma (IDC) or pure DCIS, less than or equal to 20mm maximum size.
* Lobular carcinoma in situ (LCIS) is permitted.
* Histologic grade I or II
* Estrogen receptor (ER) +/- progesterone receptor (PR) positive in greater than or equal to 10% of cells and HER2 receptor-negative.
* Tumour bed identifiable on imaging via surgical clips
* Clear surgical margins
* Sentinel nodes negative (at least one node taken if invasive and no isolated tumour cells)
* No evidence of distant metastasis

Exclusion Criteria:

* Ink on surgical margins or positive histological margins
* Lymphatic vessel invasion (LVI)
* Bilateral breast cancer
* Invasive lobular carcinoma
* Pleomorphic LCIS
* Multifocal or multicentric invasive cancer
* Invasive carcinoma with associated DCIS greater than or equal to 30mm.
* Patients receiving neoadjuvant chemotherapy, anti-HER2 agents or endocrine therapy
* Patients receiving adjuvant chemotherapy or anti-HER2 agents.
* Previous Hodgkin's lymphoma requiring mantle radiation
* Prior radiation therapy to the ipsilateral breast
* Triple-negative breast cancer
* Documented mutation of BRCA1, BRCA2 or TP53, or at high genetic risk of breast cancer
* Known inflammatory conditions associated with higher complications after RT, such as active scleroderma, systemic lupus erythematosus (requiring steroids or immune suppressive therapy)
* Oncoplastic surgery where the primary tumour site is difficult to delineate
* No previous cancer (except BCC or SCC of the skin) unless in remission beyond five years of diagnosis
* People who are pregnant or planning to become pregnant
* People who are unable or unwilling to comply with protocol requirements.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2030-07 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Patient-reported breast-related cosmetic outcome, | 36 months post randomisation
  Proportion of patients with a moderate or worse adverse cosmetic outcome, defined as a score of greater than or equal to 2.5 on the aesthetic sub-scale of the Breast Cancer Treatment Outcome Scale-12 (BCTOS-12).

SECONDARY OUTCOMES:
Patient-reported breast-related cosmetic outcome | Baseline, 8 weeks post-treatment, 6, 12, 18, 24 and 36-months post randomisation.
  BCTOS-12 aesthetic sub-scale scores
Patient-reported breast-related functional outcome | Baseline, 8 weeks post-treatment, 6, 12, 18, 24 and 36-months post randomisation.
  BCTOS-12 functional sub-scale scores
Patient-reported quality of life | Baseline, 8 weeks post-treatment, 6, 12, 18, 24 and 36-months post randomisation.
  BREAST-Q (V2.0) questionnaire scores for the following Breast Conserving Therapy (Post-operative) modules: - Physical well-being: chest - Satisfaction with breasts - Adverse effects of radiation - Fatigue - Impact on work
Ipsilateral breast tumour recurrence (IBTR) | Up to 36 months post-randomisation
  Cumulative incidence of local (true) recurrences of breast cancer within the index quadrant or newly diagnosed breast cancer within any other quadrant of the ipsilateral breast measured using results from standard of care imaging (mammogram, ultrasound, MRI).
Regional Recurrence | Up to 36 months post-randomisation
  Cumulative incidence of any recurrence in the ipsilateral axillary, supraclavicular or internal mammary chain with or without recurrence in the breast or elsewhere measured using results from standard of care imaging (mammogram, ultrasound, MRI).
Locoregional disease recurrence | Up to 36 months post-randomisation
  Cumulative incidence of IBTR plus any recurrence in the ipsilateral axillary, supraclavicular or internal mammary chain
Distant disease recurrence | Upto 36 months post-randomisation
  Cumulative incidence of metastases to distant organs or bone sites measured using results from standard of care imaging (mammogram, ultrasound, MRI).
Patterns of care for treatment of disease recurrence (IBTR, locoregional, or metastatic) | Upto 36 months post-randomisation
  Documented in patients' medical records
Patient satisfaction with treatment | At 8-weeks and 12 months post-treatment.
  Assessed qualitatively via an open-ended question: "Please write about your experience with breast cancer treatment, specifically focusing on your treatment with accelerated partial breast irradiation (APBI). Think about how you felt physically and emotionally and what the greatest challenges were during this time."

CONTACTS AND LOCATIONS:
Overall Officials: John Boyages, MB BS(Hons), FRANZCR, PhD, AM, Study Chair — Integrated Community Oncology Network
Locations (2):
- Australia (2):
  - Icon Cancer Centre Wahroonga, Wahroonga, New South Wales
  - Icon Cancer Centre Windsor Gardens, Windsor Gardens, South Australia

IPD SHARING:
Plan to Share IPD: No